CLINICAL TRIAL: NCT05332626
Title: Can Lactobacillus Acidophilus Decrease the Risk of Postmenopausal in Women?
Brief Title: Lactobacillus Acidophilus and Postmenopausal Women
Acronym: LaBon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Life Sciences (Other)
Collaborators: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Iskandar Harahap, Principal Investigator, Poznan University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 668/21
Record Dates: First submitted 2022-03-23; First posted 2022-04-18 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Bone Loss; Post Menopausal Osteoporosis; Mineralization
Keywords: Probiotic; Lactobacillus acidophilus; Calcium status; Bone resorption; Bone formation; Post Menopausal Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis, Postmenopausal; Calcinosis; Bone Resorption

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trail
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): The probiotic group will receive a supplement diet capsule consisting of Lactobacillus acidophilus UALa-01™ with a dose of 1x10^9 CFU for 12 weeks
  Interventions: Dietary Supplement: Probiotic group
- Placebo group (Placebo Comparator): The placebo group will receive a capsule that consists of the excipient (maize starch and maltodextrins) for 12 weeks
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Probiotic group — The probiotic gorup is focused on the treatment of postmenopause osteoporosis women with a capsule cointained 1x10^9 CFU of Lactobacillus acidophilus UALa-01™/day (30 people)
  Arms: Probiotic group
Dietary Supplement: Placebo group — The group is assigned on the treatment of postmenopause osteoporosis women without probiotic intervention (30 people)
  Arms: Placebo group

SUMMARY:
This study aims to evaluate the effect of Lactobacillus acidophilus supplementation on calcium status and bone densitometry in postmenopausal women in a randomized, double-blind placebo-controlled study.

DETAILED DESCRIPTION:
This study has three steps; namely, 1st step is to prepare the diet supplementation of probiotics and placebo. 2nd step is to perform the randomized, double-blind placebo-controlled clinical trial. 3rd step is to analyze the effects of L. acidophilus UALa-01™ in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 45 to 70 years old with more than one year since last menstruation;
2. Body mass index (BMI): 27.0 kg/m2 to 34.9 kg/m2;
3. All female participants who accepted bone densitometry measurement

Exclusion Criteria:

1. The secondary form of obesity, the pharmacological treatment for obesity (in the three months before the study), history of bariatric surgery;
2. Other gastrointestinal disorders, especially: inflammatory bowel diseases, celiac disease, gastritis and duodenitis, pancreatic disorders, gastrointestinal symptoms suggestive of irritable bowel syndrome;
3. Pharmacotherapy of lipid disorders or hypertension in the three months before enrollment
4. Clinically significant acute inflammatory process (elevated hsCRP)
5. Abnormal kidney function (GFR <60mL/min/1,73m2);
6. Participation in a body mass management study;
7. The use of drugs known to modify body mass or food intake;
8. Hormone replacement therapy;
9. History of following alternative diets (diets with the altered amount of macronutrients, vegan or vegetarian diets, high-fiber diet, a diet with high quantities of fermented food (>400 g/day), diet fortified with prebiotics- and probiotics-functional food, elimination diets, low-calorie diets) within three months before the study;
10. History of use of any dietary supplements, including calcium, in the three months before the study;
11. History of intake of antibiotics, probiotics, prebiotics (and synbiotics) within three months before the study;
12. Type 2 diabetes - - requiring the introduction and/or change of pharmacological treatment in the 2 years before the trial or during intervention;
13. Dyslipidemia - requiring the introduction and/or change of pharmacological treatment in the 6 months before the trial or during intervention;
14. Hypertension - requiring the introduction and/or change of pharmacological treatment in the 6 months before the trial or during intervention;
15. Another chronic pharmacotherapy: nonsteroidal anti-inflammatory drugs, proton pump inhibitors, anticoagulants, drugs causing metabolic alteration, e.g., SFAs (second-generation antipsychotics);
16. Diseases requiring nutritional requirement and chronic supplementation;
17. Alcohol (>20g/d), nicotine or drug abuse;
18. Mental disorders, including eating disorders;
19. Cancer, autoimmune diseases;
20. Any other condition that, in the opinion of the investigators, would make participation not in the best interest of the subject, or could prevent, limit, or confound the efficacy of the study any diseases, disorders, and therapies, which may influence on final results of the study or pose a risk for subjects health.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Life Sciences, Poznan, Greater Poland Voivodeship, Poland

RESULTS

PARTICIPANT FLOW:
Groups:
- Probiotic Group: Participants received a daily capsule containing Lactobacillus acidophilus UALa-01™ (1×10⁹ CFU) for 12 weeks to evaluate its effect on postmenopausal osteoporosis.
- Placebo Group: Participants received a daily placebo capsule containing maize starch and maltodextrins for 12 weeks as a control for evaluating the probiotic intervention.
Period: Overall Study
Arm/Group | Probiotic Group | Placebo Group
Started | 32 | 32
Completed | 30 | 25
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Population: Postmenopausal women aged 45-70 with a BMI of 27.0-34.9 kg/m² were recruited, meeting criteria of amenorrhea for 12+ months. Exclusions included diabetes, secondary obesity, GI diseases, recent dietary supplements, pharmacotherapy for lipid issues, smoking, alcohol/drug abuse, or recent antibiotic use. Of 64 eligible participants, 55 completed the 12-week intervention, randomized in a double-blind design to probiotic or placebo groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotic Group | Placebo Group | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (6.5) | 56.5 (5.8) | 58.1 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Poland | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Calcium
Description: measure the calcium concentration in serum and hair
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Probiotic Group | Placebo Group
Number analyzed (Participants) | 30 | 25
mmol/L | 1.88 (0.44) | 2.04 (0.09)

2. Primary Outcome: DXA
Description: bone densitometry analysis
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: g/cm2
Groups:
- Probiotic Group; Placebo Group: Measure BMD Total Body using DXA
Arm/Group | Probiotic Group | Placebo Group
Number analyzed (Participants) | 30 | 25
g/cm2 | 1.12 (0.12) | 1.15 (0.11)

3. Secondary Outcome: Body Mass
Description: measure body mass in kilograms
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Probiotics Group; Placebo Group: Measure Body Mass (kg)
Arm/Group | Probiotics Group | Placebo Group
Number analyzed (Participants) | 30 | 25
kg | 72.22 (15.21) | 73.88 (13.45)

4. Secondary Outcome: Calcium Intake
Description: assessing calcium intake with the questionnaire
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: gram
Groups:
- Probiotics Group; Placebo Group: Measure calcium intake
Arm/Group | Probiotics Group | Placebo Group
Number analyzed (Participants) | 30 | 25
gram | 1,115.81 (529.76) | 894.72 (381.84)

5. Secondary Outcome: Biomarkers of Bone Turnover: CTX
Description: measure the concentration of C-terminal telopeptide of type I collagen (CTX) in serum
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Probiotics Group; Placebo Group: measure the concentration of C-terminal telopeptide of type I collagen (CTX) in serum
Arm/Group | Probiotics Group | Placebo Group
Number analyzed (Participants) | 30 | 25
pg/ml | 5.67 (0.52) | 5.11 (0.52)

6. Secondary Outcome: Biomarkers of Bone Turnover: TRAP5b
Description: measure the concentration of tatrate-resistant acid phosphatase isoform-5b (TRAP5b) in serum
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Probiotics Group; Placebo Group: measure the concentration of tatrate-resistant acid phosphatase isoform-5b (TRAP5b) in serum
Arm/Group | Probiotics Group | Placebo Group
Number analyzed (Participants) | 30 | 25
ng/ml | 26.09 (9.31) | 21.13 (6.33)

7. Secondary Outcome: Biomarkers of Bone Resorption: BSAP
Description: measure the concentration of bone-specific alkaline phosphatase (BSAP) in serum
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Probiotics Group; Placebo Group: measure the concentration of bone-specific alkaline phosphatase (BSAP) in serum
Arm/Group | Probiotics Group | Placebo Group
Number analyzed (Participants) | 30 | 25
ng/ml | 10.90 (1.56) | 11.38 (1.96)

8. Secondary Outcome: Biomarkers of Bone Resorption: PINP
Description: measure the concentration of N-terminal propeptide of type I procollagen (PINP) in serum
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Probiotics Group; Placebo Group: measure the concentration of N-terminal propeptide of type I procollagen (PINP) in serum
Arm/Group | Probiotics Group | Placebo Group
Number analyzed (Participants) | 30 | 25
ng/ml | 2.64 (0.52) | 2.66 (0.52)

ADVERSE EVENTS:
Time Frame: 2 years
Description: All adverse events were assessed based on ClinicalTrials.gov definitions. The study population consisted of postmenopausal women receiving either a placebo or a probiotic (Lactobacillus acidophilus UALa-01™) recognized as generally safe (GRAS). No Serious Adverse Events (SAEs) or deaths were reported during the 12-week intervention. The data presented reflect all collected and assessed adverse events, regardless of their relatedness to the intervention.
Arm/Group | Probiotic Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/25
Other Adverse Events (participants affected / at risk) | 0/30 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT05332626/Prot_000.pdf